CLINICAL TRIAL: NCT00464828
Title: Internal Jugular Vein and Carotid Artery Anatomic Relation as Determined by Ultrasonography in Obstetric Patients
Brief Title: Ultrasound Imaging of Neck Blood Vessels in Pregnant and Non-Pregnant Women
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Other Study IDs: 06-04; 06-0217-E
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2007-11-15 (Estimated); Status verified 2007-11

CONDITIONS: Pregnancy
Keywords: Central venous cannulation; Internal jugular vein; Ultrasound; Obstetrics
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Internal jugular vein cannulation
Device: ultrasound

SUMMARY:
There is no data regarding success rates and incidence of carotid punctures during central venous cannulation (CVC) in the pregnant patients. We hypothesize that because of the anatomical and physiological changes associated with pregnancy, these patients are at higher risk of procedure failure and carotid puncture than the general population. The purpose of our study is to determine the success rate and incidence of carotid punctures using an ultrasound-simulated procedure in pregnant and non-pregnant patients.

DETAILED DESCRIPTION:
There is no data regarding success rates and incidence of carotid punctures during central venous cannulation (CVC) in pregnant patients. We hypothesize that because of the anatomical and physiological changes associated with pregnancy, these patients are at higher risk of procedure failure and carotid puncture than the general population. The purpose of our study is to determine the success rate and incidence of carotid punctures using an ultrasound-simulated procedure in pregnant and non-pregnant patients.

Pregnant patients and adult female volunteers (controls) were recruited. Subjects were placed supine with wedge under the right hip, and head turned 35 degrees to the left. Two different approaches for CVC, the central landmark and the palpatory approach were used. The ease of identification of the landmarks was noted. CVC was simulated using an ultrasound probe, on pre-marked points. Ultrasound images were obtained, within the same parasagittal plane, directed 30 degrees caudad, in a manner simulating how a syringe and needle would be placed for central venous cannulation. The investigator placing the probe was blinded to the image being generated. The vertical cursor of the ultrasound, which serves to delineate the path of a needle, was placed in the image. If the cursor intersects the vein, the attempt is considered successful. If the first attempt is not successful, the investigator placing the probe was asked to redirect the probe to the second and if necessary to the third marked point. This was done for each approach. If the cursor intersects the carotid artery, the attempt is considered an accident and no further attempts were made. In addition to determining the success rate and the incidence of carotid punctures, the relative position of vein and artery was studied in each patient. For each approach, the best image was recorded, and three experienced anesthesiologist scored the images for vein and artery degree of overlapping.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients
* Healthy non-pregnant female volunteers

Exclusion Criteria:

* Urgent, emergent or hemodynamically unstable patients
* Patients with known abnormal neck anatomy, previous surgery or trauma involving the neck, or prior cannulation of neck vessels

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2006-11; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD PhD, Principal Investigator — Mount Sinai Hosiptal
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Siddiqui N, Goldszmidt E, Haque SU, Carvalho JC. Ultrasound simulation of internal jugular vein cannulation in pregnant and non-pregnant women. Can J Anaesth. 2010 Nov;57(11):966-72. doi: 10.1007/s12630-010-9374-5. Epub 2010 Sep 10. PMID 20830543